CLINICAL TRIAL: NCT05172141
Title: A Safety, Tolerability, and Efficacy Study of IBI314 in Patients With Mild to Moderate COVID-19
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Due to the company's development strategy adjustment, Innovant Biologics decided not to continue this study after consultation with investigators.
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CIBI314B201
Record Dates: First submitted 2021-12-24; First posted 2021-12-29 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — P5-22 and P14-44 drug combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Masking participant and Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IBI314 (Experimental): Low/medium/high dose, intravenously, once, on Day 1
  Interventions: Biological: IBI314(low dose); Biological: IBI314(high dose); Biological: IBI314(medium dose)
- Placebo (Placebo Comparator): Placebo, intravenously, once, on Day 1
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: IBI314(low dose) — intravenously, once, on Day 1
  Arms: IBI314
Biological: IBI314(high dose) — intravenously, once, on Day 1
  Arms: IBI314
Biological: IBI314(medium dose) — intravenously, once, on Day 1
  Arms: IBI314
Other: Placebo — intravenously, once, on Day 1
  Arms: Placebo

SUMMARY:
This is a Phase 1/2 study evaluating the safety, tolerability and efficacy of IBI314.

DETAILED DESCRIPTION:
Phase 1 is a randomized, double-blind, placebo-controlled, single ascending dose study in up to 24 health volunteers. This phase of the study is designed to assess the safety, tolerability and PK of IBI314 administered as a single IV infusion. Phase 2 is a randomized, double-blind, placebo-controlled expansion study in approximately 198 mild to moderate adult patients with COVID-19. This phase of the study is designed to assess the efficacy, safety, PK and PD of IBI314.

ELIGIBILITY:
Main Inclusion Criteria:

First onset of COVID-19 symptoms <7 days at randomization, symptoms such as fever and/or chills, fatigue, muscle or body aches, headache, new loss of taste or smell, sore throat, congestion or runny nose, nausea or vomiting, and diarrhea.

Have a positive SARS-CoV-2 Reverse Transcription-Polymerase Chain Reaction (RT-PCR) test using an appropriate sample such as nasopharyngeal (NP), nasal, oropharyngeal, or saliva within 72 hours prior to randomization. A historical record of a positive result from a test conducted ≤72 hours prior to randomization is acceptable.

Male or female patients ≥18 years of age at the time of signing informed consent.

Agree to use an adequate method of contraception throughout the study period and for 6 months after the dose of study drug is administered.

Women of childbearing potential (WOCBP) must have a negative urinary pregnancy test at screening.

Main Exclusion Criteria:

Have oxygen saturation (SpO2) ≤93 % on room air at sea level or a ratio of arterial oxygen partial pressure (PaO2 in millimeters of mercury) to fractional inspired oxygen (FiO2) <300, respiratory rate ≥30 per minute, heart rate ≥125 per minute.

Have evidence of multi-organ dysfunction/failure. Systolic blood pressure <90 mmHg, diastolic blood pressure <60 mmHg, or requiring vasopressors.

Require or anticipated impending need for endotracheal intubation, mechanical ventilation, oxygen delivered by high-flow nasal cannula noninvasive positive pressure ventilation, extracorporeal membrane oxygenation (ECMO).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 222 (Actual)
Dates: Start 2021-12-31 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Number of treatment related AEs | 29 days after the last participant is randomized
  Any AEs and SAEs occurring during the study
Virologic efficacy Evaluation | 7 days after the last participant is randomized
  Time-weighted average change in viral shedding from baseline through Day 7 as measured by RT-qPCR in NP swab samples

SECONDARY OUTCOMES:
maximum concentration (Cmax) | 29 days after the last participant is randomized
  PK parameters to be evaluated for IBI314 including maximum concentration (Cmax) will be determined when appropriate.
area under the concentration-time curve (AUC) | 29 days after the last participant is randomized
  PK parameters to be evaluated for IBI314 including area under the concentration-time curve (AUC) will be determined when appropriate.
half-life (t1/2) | 29 days after the last participant is randomized
  PK parameters to be evaluated for IBI314 including half-life (t1/2) will be determined when appropriate.
clearance (CL) | 29 days after the last participant is randomized
  PK parameters to be evaluated for IBI314 including clearance (CL) will be determined when appropriate.
volume of distribution (V) | 29 days after the last participant is randomized
  PK parameters to be evaluated for IBI314 including volume of distribution (V) will be determined when appropriate.
The incidence of anti-IBI314 antibody (ADA) and neutralizing antibody (NAb) in serum before and after study drug administration | 29 days after the last participant is randomized
  Each patient will be tested for anti-drug (IBI314) antibody (ADA), and ADA-positive serum samples will continue to be tested for neutralizing antibodies (NAb).
Time to alleviation of symptoms (going to mild or absent) | 29 days after the last participant is randomized
  This is a clinical efficacy outcome measure.
Proportion of patients with all-cause mortality by Day 29 | 29 days after the last participant is randomized
  This is a clinical efficacy outcome measure.
Time to negative RT-qPCR in NP swab samples with no subsequent positive RT-qPCR | 29 days after the last participant is randomized
  This is a virologic efficacy outcome measure.
Change from baseline in viral shedding on Day 7, 11, 22 | 7, 11, 22 days after the last participant is randomized
  This is a virologic efficacy outcome measure.
Time-weighted average change in viral shedding from baseline through D11 as measured by RT-qPCR in NP swab samples | 11 days after the last participant is randomized
  This is a virologic efficacy outcome measure.
Time-weighted average change in viral shedding from baseline through D22 as measured by RT-qPCR in NP swab samples. | 22 days after the last participant is randomized
  This is a virologic efficacy outcome measure.
Proportion of patients demonstrating symptoms alleviation on D3, 7, 15, 22, 29 | 3, 7, 15, 22, 29 days after the last participant is randomized
  This is a clinical efficacy outcome measure.
Proportion of patients who become severe COVID-19 by Day 29 | 29 days after the last participant is randomized
  This is a clinical efficacy outcome measure.
Proportion of patients requiring mechanical ventilation by day 29 | 29 days after the last participant is randomized
  This is a clinical efficacy outcome measure.

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No